CLINICAL TRIAL: NCT02385032
Title: Comparative Bioavailability Study of UDCA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DW_UDCA001
Record Dates: First submitted 2015-03-04; First posted 2015-03-11 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
MeSH Terms: interventions — Ursodeoxycholic Acid

ARMS (2):
- AB (Experimental): Ursodiol followed by URSO Forte
  Interventions: Drug: Ursodiol; Drug: URSO Forte
- BA (Experimental): URSO Forte followed by Ursodiol
  Interventions: Drug: Ursodiol; Drug: URSO Forte

INTERVENTIONS:
Drug: Ursodiol
Drug: URSO Forte

SUMMARY:
The purpose of this study is to evaluate bioavailability of two formulations of ursodiol.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 19.0 and ≤ 30.0 kg/m2.
* No clinically significant findings in a 12-lead electrocardiogram (ECG)
* Be informed of the nature of the study and give written consent prior to any study procedure

Exclusion Criteria:

* Known history or presence of any clinically significant medical condition
* Participated in a clinical trial which involved administration of an investigational medicinal product within 30 days prior to drug administration, or recently participated in a clinical investigation that, in the opinion of the investigator, would jeopardize subject safety or the integrity of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
AUClast | 72 hours
Cmax | 72 hours